CLINICAL TRIAL: NCT03621787
Title: Assessing the Safety and Efficacy of the SubQ Assist Implant Insertion Device
Brief Title: Assessing the Safety and Efficacy of a Novel Subcutaneous Implant Insertion Device on Healthy Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Expiration of study funds.
Sponsor: University of Michigan (Other)
Collaborators: Michigan Translation and Commercialization for Life Sciences Hub (Other); Grand Challenges Canada (Other); VentureWell (Industry); Unite for Sight (Other)
Responsible Party: Principal Investigator, Ibrahim Mohedas, Postdoctoral Fellow, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SubQAssist0001
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Participants in trial will be within a single study arm. All participants will have a placebo subcutaneous implant inserted with the device being studied. The implant accuracy will be assess through palpation and ultrasound depth measurements. The implant will then be removed. Safety will be assessed by measuring bruising, bleeding, and pain to participant. A follow-up questionnaire will assess pain, bruising, and infection risk. A final visit will assess pain, bruising, and infection risk by a physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single arm study: implant insertion (Experimental): Participants in trial will be within a single study arm. All participants will have a placebo subcutaneous implant inserted with the device being studied. The implant accuracy will be assess through palpation and ultrasound depth measurements. The implant will then be removed. Safety will be assessed by measuring bruising and bleeding. A follow-up questionnaire will assess bruising and infection risk. A final visit will assess bruising and infection risk by a physician.
  Interventions: Device: Implant insertion device

INTERVENTIONS:
Device: Implant insertion device — Device designed to assist healthcare providers in administering subcutaneous implants safely and accurately.
  Other Names: SubQ Assist

SUMMARY:
The investigators have created a device designed to make it easier to insert pharmaceutical implants under the skin. The device uses a blood pressure cuff to hold the skin on a person's arm in place while a mechanical guide places implants underneath the skin. This device may prevent implants from being embedded too deeply.

The investigators are performing this study to determine the safety and efficacy of the device for use in adult women. The study will determine if the implants are placed accurately under the skin (in the sub-dermal layer). It will also assess if the device causes any discomfort or last pain from use.

DETAILED DESCRIPTION:
Subcutaneous contraceptive implants are one of the preferred methods of long-term contraception by the World health Organization and ministries of health in low- and middle-income countries. These implants offer between three and five years of protection (allowing women to safely space pregnancies and thereby reduce maternal and infant mortality), are 99.95% efficacious, allow women to return to fertility quickly when removed, requires no daily/monthly effort on the part of the woman, and cause minimal side effects in comparison to other methods. However, availability of contraceptive implants in rural areas is limited due to the skill necessary to administer them safely and accurately.

The investigators have created a device designed to make it easier to insert pharmaceutical implants under the skin. The device uses a blood pressure cuff to hold the skin on a person's arm in place while a mechanical guide places implants underneath the skin. This device is designed to prevent implants from being embedded too deeply.

In this trial, the investigators will use the implant insertion device with a placebo sub-cutaneous implant. Implants will be inserted with the device and the accuracy of the placement will be assessed through palpation and ultrasound depth measurements. This data will allow the investigators to assess whether the device ensures accurate insertions of sub-cutaneous implants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects aged 18 to 49
* Ability to understand study procedure and informed consent document

Exclusion Criteria:

* Patients with a history of keloid scarring
* Pregnancy
* Any rashes or skin conditions around the insertion site
* Known silicone allergies
* Known allergy to lidocaine
* History of bleeding disorders or abnormal bleeding

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen H Sienko, PhD, Principal Investigator — Associate Professor; Carrie L Bell, MD, Principal Investigator — Assistant Professor
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm Study: Implant Insertion
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study: Implant Insertion
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9
Arm circumference [Mean (Standard Deviation); unit: centimeters] — Arm circumference measurement taken at the epicondyle in centimeters
  centimeters | 23.67 (1.95)
Weight [Mean (Standard Deviation); unit: kilograms] | 62.57 (11.86)
Height [Mean (Standard Deviation); unit: centimeters] | 167.5 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Implant Depth: Distal End
Description: Depth of distal end of implant beneath the skin after insertion. Measured via high frequency ultrasound with linear probe. Measured in centimeters below skin surface. Measurements will be aggregated via mean and standard deviation.
Time Frame: Up to 60 minutes after insertion
Measure: Mean (Standard Deviation); unit: centimeters
Units Other Than Participants: Implants
Arm/Group | Single Arm Study: Implant Insertion
Number analyzed (Participants) | 9
Number analyzed (Implants) | 18
centimeters | 0.26 (0.05)

2. Primary Outcome: Implant Depth: Proximal End
Description: as for outcome 1
Time Frame: Up to 60 minutes after insertion
Measure: Mean (Standard Deviation); unit: centimeters
Units Other Than Participants: implants
Arm/Group | Single Arm Study: Implant Insertion
Number analyzed (Participants) | 9
Number analyzed (implants) | 18
centimeters | .35 (.07)

3. Primary Outcome: Implant Palpability
Description: A binary (yes/no) assessment of whether the implant is palpable by a physician under the skin after insertion. Measurements will be aggregated based on percent of implants that are palpable.
Time Frame: Up to 15 minutes after insertion
Measure: Number; unit: palpable implants
Units Other Than Participants: implants
Arm/Group | Single Arm Study: Implant Insertion
Number analyzed (Participants) | 9
Number analyzed (implants) | 18
palpable implants | 18

4. Secondary Outcome: Number of Participants With Bruising
Description: Bruising may occur from inflation of the blood pressure cuff over the device being studied. A binary assessment of bruising (yes/no) will be assessed by the physician after insertion.
Time Frame: Up to 15 minutes after insertion.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study: Implant Insertion
Number analyzed (Participants) | 9
Participants | 1

5. Secondary Outcome: Presence of Bruising
Description: Bruising may occur from inflation of the blood pressure cuff over the device being studied. Bruising will be assessed by the participant in a survey (binary yes/no indication of bruising around insertion site).
Time Frame: 7 to 14 days after insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study: Implant Insertion
Number analyzed (Participants) | 9
Participants | 1

6. Secondary Outcome: Number of Participants With More Bleeding Than Typical
Description: Bleeding from insertion will be assessed by the physician who has extensive training with implant insertions. The number of participants with more bleeding than is typically associated with insertion will be measured.
Time Frame: Up to 10 minutes after insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study: Implant Insertion
Number analyzed (Participants) | 9
Participants | 1

7. Secondary Outcome: Number of Participants With Signs of Infection
Description: Infection will be assessed during the follow-up questionnaire. A binary assessment (yes/no) of the following will be assessed by the participant. 1) Is there currently any fluid draining from the incision? 2) Is there currently any redness or swelling of the insertion site? 3) Is there currently any bleeding from the insertion site?
  Participants who answer "Yes" to all three questions are deemed to have shown signs of infection.
Time Frame: 7 to 10 days after insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study: Implant Insertion
Number analyzed (Participants) | 9
Participants | 0

8. Secondary Outcome: Number of Participants With Signs of Infection
Description: A follow-up appointment with all participants was conducted by the physician who administered the implant. A binary assessment (yes/no) of the following will be assessed for each participant by the physician. 1) Is there currently any fluid draining from the incision? 2) Is there currently any redness or swelling of the insertion site? 3) Is there currently any bleeding from the insertion site?
  If the physician answers "Yes" to all three questions, the participant is deemed to have shown signs of infection.
Time Frame: 21 to 28 days after insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study: Implant Insertion
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were tracked for each participant from the beginning of the study through their follow-up appointment. Up to 28 days.
Arm/Group | Single Arm Study: Implant Insertion
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study: Implant Insertion (N=9)
Difficulty removing implant (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-11-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT03621787/Prot_001.pdf